CLINICAL TRIAL: NCT06947473
Title: Single Center, Open Label, Non Randomized, Single Arm Clinical Study of Cord Blood CD19-BCMA CART Cell Therapy for Refractory Lupus Nephritis (SLE-LN), Systemic Sclerosis (SSc), and Primary Sjogren's Syndrome With Pulmonary Hypertension (pSS PAH)
Brief Title: Umbilical Cord Blood CD19-BCMA CART Cell Therapy for SLE-LN, SSc, andpSS PAH.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of the department of Immunotherapy for Hematopoietic Malignancies, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2025-025
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-05

CONDITIONS: Refractory Lupus Nephritis; Systemic Sclerosis; Primary Sjogren's Syndrome Combined With Pulmonary Hypertension
MeSH Terms: conditions — Lupus Nephritis; Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- umbilical cord blood CD19-BCMA CAR T cell therapy. (Experimental): Patients were treated with umbilical cord blood CD19-BCMA CAR T cell therapy.
  Interventions: Drug: umbilical cord blood CD19-BCMA CAR-T cells infusion

INTERVENTIONS:
Drug: umbilical cord blood CD19-BCMA CAR-T cells infusion — Approximately 3-5 days prior to umbilical cord blood CD19-BCMA CAR-T cell infusion, subjects are treated with FC regimen (fludarabine and cyclophosphamide) for lymphodepletion. CAR-T cell infusion are performed 48 h after completion of chemotherapy.

SUMMARY:
This is a single-center, open-label, non-randomized, single-arm clinical trial. Patients with refractory lupus neritis (SLE-LN), systemic sclerosis (SSc), and primary Sjogren syndrome combined with pulmonary artery hypertension (pSS-PAH receive umbilical cord blood CD19-BCMA CAR T cell therapy. The primary objective is to prospectively assess the safety of umbilical cord blood CD19BCMA CAR T cell therapy in patients with refractory lupus nephritis (SLE-LN), systemic sclerosis (SSc), and primaryjogren syndrome combined with pulmonary artery hypertension. The primary endpoint is the type and incidence of dose-limiting toxicity (DLT) within 28 days after theusion of umbilical cord blood CD19-BCMA CAR T cells. It is anticipated that 45-54 participants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* 1. Refractory lupus nephritis (LN):

According to the 2019 American College of Rheumatology (ACR) criteria and the 2018 International Society of Nephrology (ISN)/Society of Nephrology (RPS) criteria (see Appendix 3), confirmed by renal tissue biopsy as active, proliferative lupus nephritis, type III or IV [excluding type III (C), IV-S (C), and IV-G (C)], or type III/IV combined with type V. Biopsy must be performed within 6 months prior to the screening visit or during the screening period.

1. Male or female patients aged 3-65 years old;
2. Systemic lupus erythematosus that meets the 2019 American College of Rheumatology (ACR)/European Union of Rheumatology Associations (EULAR) classification criteria (see Annex 5);
3. The result of the anti nuclear antibody (ANA) test is clearly positive, that is, the ANA titer is ≥ 1:80 (equivalent test result based on Hep-2 immunofluorescence detection method or enzyme immunoassay method), and/or at the screening visit, the anti dsDNA serum antibody test is positive (≥ 30 IU/mL based on ELISA detection method) according to the test results of the research center laboratory.
4. B cell CD19+expression and discontinuation of immunosuppressive agents for more than 1 week;
5. No severe allergic constitution;
6. Physical condition score (ECOG) 0-2 points;
7. Expected survival period ≥ 90 days;
8. The subjects and/or their guardians are able to understand and willing to sign a written informed consent form; 2. Systemic sclerosis (SSc):

<!-- -->

1. The selected patient or their legal representative voluntarily signs the informed consent form.
2. Age range: 6-65 years old (including 6 and 65 years old), gender is not limited.
3. According to the SSc classification criteria proposed by the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) in 2013, the highest score under the same item, ≥ 9 points, can be classified as SSc (Attachment 6).
4. Or if one sufficient condition is met, that is, the skin of both fingers thickens and extends to the proximal end of the metacarpophalangeal joint, it can be directly classified as SSc.

3. Primary Sjogren's syndrome with pulmonary hypertension (pSS PAH):

(1) The selected patients or their legal representatives voluntarily sign informed consent.

(2) Age range: 18-65 years old (including 18 and 65 years old), gender is not limited.

(3) Patients with refractory connective tissue disease (pulmonary arterial hypertension):

1. Diagnosed with primary Sjogren's syndrome according to the 2002 AECG classification criteria or the 2016 ACR/EULAR classification criteria
2. Confirmed by right heart catheterization to meet the diagnostic criteria for PAH (as defined in the 2022 ESC/ERS guidelines for the diagnosis and treatment of pulmonary arterial hypertension):

   * Resting mean pulmonary artery pressure (mPAP) ≥ 20mmHg;

     * Pulmonary artery wedge pressure (PAWP) ≤ 15mmHg;

       ③ Resting pulmonary vascular resistance (PVR)>2WU; (4) PAH did not reach the risk stratification of low-risk group patients. Low risk patients need to meet: ① WHO heart function classification I-II; ② 6-minute walking distance (6MWD)>440 meters; ③ BNP<50ng/L， Or NT proBNP<300ng/L; ④ Right atrial pressure (RAP)<8mmHg and cardiac index (CI) ≥ 2.5 L · min-1 · m-2.

       (5) Prior to the first administration of the investigational drug, a stable dose of standard treatment was received, including corticosteroids (prednisone 0-30mg/day, or equivalent other formulations) for at least 4 weeks; Antimalarial drugs and monotherapy immunosuppressants (allowed immunosuppressants are limited to: mycophenolate mofetil or mycophenolate mofetil ≤ 1.5g/day, azathioprine or 6-mercaptopurine ≤ 2mg/kg/day, methotrexate ≤ 15mg/week, leflunomide ≤ 20mg/day) should be used for at least 12 weeks, and should not be increased or replaced within 24 weeks after drug treatment. Prior to drug treatment, use PAH targeted drugs of less than three types (including prostaglandin analogs, endothelin receptor antagonists, PDE-5 inhibitors, and guanylate cyclase agonists), which have been stable for at least 4 weeks and have not been increased or replaced within 24 weeks after drug treatment.

       (6) Clinicians assess the patient's condition and allow the use of corticosteroids at a dose not exceeding 10mg prednisone or its equivalent during the study period, and allow the discontinuation of all immunosuppressants (excluding hydroxychloroquine).

       (7) Women of childbearing age have a negative blood pregnancy test within 7 days prior to the pre-treatment treatment; Any male and female patient with fertility must agree to use an effective contraceptive method throughout the entire study process and for at least one year through the infusion of cell injection. The patient's fertility refers to their biological ability to give birth to live infants and have normal sexual activity. Female patients who are infertile (i.e. meet at least one of the following criteria): have undergone hysterectomy or bilateral oophorectomy, or have been medically confirmed to have ovarian failure, or have been medically confirmed to be postmenopausal (with at least 12 consecutive months of amenorrhea without pathological or physiological reasons).

       (8) Having appropriate organ function, it must meet the following standards: Aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal (ULN); Alanine aminotransferase (ALT) ≤ 3 times ULN; Total serum bilirubin ≤ 2 times ULN, unless the patient has a record of Gilbert syndrome; Bilirubin ≤ 3.0 times ULN and direct bilirubin Gilbert syndrome patients with hemoglobin ≤ 1.5 times ULN can be included; There must be a minimum level of lung reserve, with oxygen saturation greater than 95% in non oxygenated state.

Exclusion Criteria:

* 1. Refractory lupus nephritis (LN):

  1) Intracranial hypertension or cerebral consciousness disorders; 2) Symptomatic heart failure or severe arrhythmia; 3) Symptoms of severe respiratory failure; 4) Accompanied by other types of malignant tumors; 5) Diffuse intravascular coagulation; 6) Suffering from sepsis or other difficult to control infections; 7) Have uncontrollable diabetes and other endocrine diseases; 8) Serious mental disorder; 9) Head MRI examination shows obvious lesions in the skull; 10) Received organ transplantation (excluding bone marrow transplantation); 11) Female patients (those with fertility) have a positive HCG test in their blood; 12) Hepatitis (including hepatitis B and C), AIDS and syphilis screening positive persons; 13）eGFR CKD-EPI < 30 ml/min/1.73m^2； 14) Any active skin disease that may interfere with the evaluation of systemic lupus erythematosus research,Including but not limited to psoriasis, dermatomyositis, systemic sclerosis, and non systemic diseases Skin manifestations of lupus erythematosus (such as skin vascular disease, pericapillary dilation)Zhang, fingertip sclerosis, rheumatoid nodules, erythema multiforme, leg ulcers)Or drug-induced lupus.

  15) Subjects who were not successfully matched during the screening period; 16) Previously received CART treatment other than CD19-CART. 2. Primary Sjogren's syndrome with pulmonary hypertension (pSS PAH):

  1) PH caused by other reasons: portal hypertension, hereditary hemorrhagic telangiectasia, etc; Congenital heart disease; Suspicious drugs and toxins; Chronic hypoxic disease-related pulmonary hypertension: moderate or severe obstructive pulmonary disease: FEV1<55%； Moderate or severe restrictive lung disease: TLC<60%； Chronic thromboembolic disease pulmonary hypertension: Pulmonary ventilation/perfusion imaging suggests moderate to high suspicion of pulmonary thromboembolism; 2) Suffering from severe active central nervous system (CNS) lupus, including seizures, psychosis, cerebrovascular accidents, or CNS vasculitis requiring therapeutic intervention within 60 days after baseline; 3) Dialysis patients or creatinine clearance rate less than 30mL/min; 4) Pregnancy or breastfeeding; 5) Merge active infections (such as sepsis, bacteremia, mycosis, uncontrolled pulmonary infections, and active tuberculosis); 6) Hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg) are positive; Hepatitis B e antibody (HBe Ab) and/or hepatitis B core antibody (HBc Ab) are positive, and the number of HBV-DNA copies is greater than the measurable lower limit; Hepatitis C (HCV) antibody positive; Positive for human immunodeficiency virus (HIV) antibodies; Individuals who test positive for syphilis antibody (TP Ab); 7) Having undergone major surgeries evaluated by researchers as unsuitable for inclusion within the previous 4 weeks prior to screening; 8) Subjects who were not successfully matched during the screening period; 9) Previously received CART treatment other than CD19-CART. 3.Systemic sclerosis (SSc)：

  1) Overlapping connective tissue diseases; Rheumatoid arthritis, systemic lupus erythematosus, or inflammatory myopathy 2) The clinical manifestations can be explained by similar diseases of SSc, such as nephrogenic systemic fibrosis, generalized scleroplakia, eosinophilic fasciitis, diabetes scleroma, scleromyedema, erythematous acrodynia, porphyria, sclerotic lichen, graft-versus-host disease, diabetes and other endocrine diseases related hand joint diseases.

  3) Suffering from severe active central nervous system (CNS) lupus, including seizures, psychosis, cerebrovascular accidents, or CNS vasculitis requiring therapeutic intervention within 60 days after baseline; 4) Dialysis patients or creatinine clearance rate less than 30mL/min; 5) Pregnancy or breastfeeding; 6) Merge active infections (such as sepsis, bacteremia, mycosis, uncontrolled pulmonary infections, and active tuberculosis); 7) Hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg) are positive; Hepatitis B e antibody (HBe Ab) and/or hepatitis B core antibody (HBc Ab) are positive, and the number of HBV-DNA copies is greater than the measurable lower limit; Hepatitis C (HCV) antibody positive; Positive for human immunodeficiency virus (HIV) antibodies; Individuals who test positive for syphilis antibody (TP Ab); 8) Having undergone major surgeries evaluated by researchers as unsuitable for inclusion within the previous 4 weeks prior to screening; 9) Subjects who were not successfully matched during the screening period; 10) Previously received CART treatment other than CD19-CART.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-18 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days
  Incidence and type of dose-limiting toxicity(DLT) within 28 days of umbilical cord blood CD19-BCMA CAR-T infusion.
Adverse events (AEs） | 30 days
  Total number, incidence and severity of adverse events (AEs) within 30 days of umbilical cord blood CD19-BCMA CAR-T infusion

SECONDARY OUTCOMES:
Overall remission rate (ORR) | 90,120 days
  The assessment of ORR by dose group at 90 and 120 Days after umbilical cord blood CD19-BCMA CAR T infusion.
Serious adverse event（SAE) | from 30 days to 2 years
  The incidence and grade of serious adverse events (SAEs) from 30 days to 2 years post-infusion

IPD SHARING:
Plan to Share IPD: Undecided